CLINICAL TRIAL: NCT03695250
Title: Phase I/II Trial of BMS-986205 and Nivolumab as First or Second Line Therapy in Hepatocellular Carcinoma
Brief Title: BMS-986205 and Nivolumab as First or Second Line Therapy in Treating Patients With Liver Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding source decision to terminate study.
Sponsor: Edward Kim (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Edward Kim, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1229924; NCI-2018-02009 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#276 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Hepatocellular Carcinoma; Stage III Hepatocellular Carcinoma AJCC v8; Stage IIIA Hepatocellular Carcinoma AJCC v8; Stage IIIB Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8; Stage IVB Hepatocellular Carcinoma AJCC v8; Unresectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — linrodostat; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (BMS-986205 and nivolumab) (Experimental): Patients receive IDO1 inhibitor BMS-986205 PO QD on days 1-14 and nivolumab IV over 30 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: IDO1 Inhibitor BMS-986205; Biological: Nivolumab

INTERVENTIONS:
Drug: IDO1 Inhibitor BMS-986205 — Given PO
  Other Names: BMS 986205; BMS-986205; BMS986205; IDO-1 Inhibitor BMS-986205; Indoleamine-pyrrole 2,3-Dioxygenase Inhibitor BMS-986205; ONO-7701
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase I/II trial studies the side effects and best dose of IDO1 inhibitor BMS-986205 (BMS-986205) when given together with nivolumab and how well it works as first or second line therapy in treating patients with liver cancer. BMS-986205 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread. Giving BMS-986205 and nivolumab may work better in treating patients with liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain the safety and tolerability of BMS-986205 in combination with nivolumab in unresectable / metastatic hepatocellular carcinoma (HCC) in the first or second line setting using Common Terminology Criteria for Adverse Events (CTCAE) version (V)5.0 criteria.

II. To determine efficacy as defined by objective response rate (ORR) of BMS-986205 in combination with nivolumab in unresectable / metastatic HCC in the first or second line setting using Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1).

SECONDARY OBJECTIVES:

I. To determine disease control rate (DCR), duration of response (DOR), progression free survival (PFS), and overall survival (OS) by RECIST 1.1 and ORR using immune RECIST (iRECIST) of BMS-986205 in combination with nivolumab in unresectable HCC. (Phase II) II. To further evaluate safety of BMS-986205 in combination with nivolumab in unresectable HCC. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of IDO1 inhibitor BMS-986205 followed by a phase II study.

Patients receive IDO1 inhibitor BMS-986205 orally (PO) once daily (QD) on days 1-14 and nivolumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 100 days, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for the trial
* Life expectancy > 12 weeks
* Histologically or imaging confirmed hepatocellular carcinoma (mixed hepatocellular/cholangiocarcinoma or fibrolamellar subtypes are excluded)
* Have disease that is not amenable for curative treatment approach
* Have measurable disease based on RECIST v1.1
* >= 1 liver lesions accessible for core biopsy that was either not previously treated by liver-directed therapy or progressed following liver-directed therapy
* Child-Pugh score of A
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count (ANC) >= 1000 cell/mm^3
* Platelet count >= 50,000/mm^3
* Hemoglobin (Hgb) >= 8 g/dL
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) =< 5 x upper limit of normal (ULN)
* Total bilirubin =< 2 ULN
* Creatinine =< 2 x ULN
* Subjects with active hepatitis B virus (hep B) are allowed if antiviral therapy for hepatitis B has been given for > 8 weeks and viral load is < 100 IU/ml prior to first dose of trial treatment. Subjects with untreated hepatitis C virus (HCV) are allowed
* Willingness to undergo mandatory pre-treatment biopsy (unless there is adequate archival tumor specimen available) and mandatory on-treatment biopsy
* Female subject of child-bearing potential must have a negative urine pregnancy =< 24 hour (hr) prior to planned treatment initiation. Women with childbearing potential and males must be willing to use adequate birth control on trial and until 5 months for women or 7 months for men after the last of study therapy
* Ability to adhere to the study visit schedule and other protocol requirements
* Participants must be able to swallow pills intact

Exclusion Criteria:

* Received more than 1 prior systemic HCC-related therapy or currently receiving HCC-related systemic treatment or participating in a clinical trial and receiving study therapy
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Known diagnosis of immunodeficiency or active autoimmune disease or requiring systemic steroid equivalent of prednisone >= 10 mg/day or any immunosuppressive therapies =< 7 days of before the first dose of the study
* Active bacterial, viral (except hepatitis B and C), or fungal infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, anti-viral therapy, anti-fungal therapy, and/or other treatment
* Active pneumonitis or history of interstitial lung disease (ILD) / pneumonitis requiring steroids
* Clinically significant ascites
* Hepatic encephalopathy
* Any significant medical condition including additional malignancies, laboratory abnormalities, or psychiatric illness that would prevent the subject from participating and adhering to study related procedures
* Live attenuated vaccine =< 30 days before the first dose of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
* Use of strong inhibitor / inducer of CYP3A4 or CYP1A2
* Known history of surgery or medical condition that may affect drug absorption, per investigator descretion
* Participants with a history of G6PD deficiency or other congenital or autoimmune hemolytic disorders. All participants will be screened for G6PD deficiency prior to enrollment using quantitative or qualitative G6PD assay results to suggest underlying G6PD deficiency
* Participants with a personal or family (i.e., in a first-degree relative) history or presence of cytochrome b5 reductase deficiency (previously called methemoglobin reductase deficiency) or other diseases that puts them at risk of methemoglobinemia. All participants will be screened for methemoglobin levels prior to enrollment using blood methemoglobin > ULN, assessed in an arterial or venous blood sample or by co oximetry
* Subjects with screening corrected QT (QTc) interval > 480 ms
* Liver directed therapy =< 4 weeks before the first dose of study
* History of esophageal or gastric variceal bleeding within 3 months of study enrollment
* Treatment with botanical preparations (e.g., herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to enrollment
* Prior history of serotonin syndrome
* Prior treatment with BMS-986205 or any other IDO1 inhibitors.
* Women who are breastfeeding
* History or presence of hypersensitivity or idiosyncratic reaction to methylene blue
* History of allergy or hypersensitivity to any study treatment components, specifically to that of BMS-986205
* Participants who have had major surgery requiring general anesthesia or significant trauma who have not recovered per physician determination for at least 14 days prior to enrollment
* Participants who have had major surgery requiring general anesthesia or significant trauma who have not recovered per physician determination for at least 14 days prior to enrollment
* Participants with uncontrolled adrenal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Kim, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (BMS-986205 and Nivolumab): Patients receive IDO1 inhibitor BMS-986205 PO QD on days 1-14 and nivolumab IV over 30 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  IDO1 Inhibitor BMS-986205: Given PO Nivolumab: Given IV
Period: Overall Study
Arm/Group | Treatment (BMS-986205 and Nivolumab)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (BMS-986205 and Nivolumab)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AE)
Description: Number of participants with adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0
Time Frame: Up to 2 years.
Measure: Number; unit: participants
Arm/Group | Treatment (BMS-986205 and Nivolumab)
Number analyzed (Participants) | 8
participants
  Diarrhea | 2
  Oral pain | 1
  Flatulence | 1
  Pruritus | 1
  Fatigue | 1
  Dyspnea | 1
  Maculopapular rash | 2
  Alk phos increased | 2
  AST increased | 3
  ALT increased | 3
  Musculoskeletal pain | 1
  Anorexia | 1
  Malaise | 1
  TSH elevation | 1
  Abdominal pain | 1
  Hyperglycemia | 1
  Pancreatitis | 1

2. Primary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to approximately 2 years, 1 month.
Measure: Number (95% Confidence Interval); unit: percentage of participans
Arm/Group | Treatment (BMS-986205 and Nivolumab)
Number analyzed (Participants) | 8
percentage of participans | 12.5 [0.3 to 52.7]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of patients that achieve an objective tumor response or have stable disease to therapy. The DCR will be estimated as the proportion of participants who experience an objective response, along with its exact 95% confidence interval.
Time Frame: Up to 2.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (BMS-986205 and Nivolumab)
Number analyzed (Participants) | 8
percentage of participants | 50 [15.7 to 84.3]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions>
Time Frame: From date of enrollment to time of progression or death, whichever occurs first, assessed up to 2.5 years
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Treatment (BMS-986205 and Nivolumab)
Number analyzed (Participants) | 8
Weeks | 8.5 [4.8 to NA] — Insufficient number of participants with events.

5. Secondary Outcome: Duration of Response (DOR)
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: From the time measurement criteria are met for CR or PR (whichever status is recorded first) until the first date that recurrence or progressive disease (PD) is objectively documented, assessed up to 2.5 years
Population: End timepoints of response were not collected from any participants to assess this outcome measure.
Arm/Group | Treatment (BMS-986205 and Nivolumab)
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival (OS)
Description: OS will be analyzed using Kaplan-Meier methods; medians and 95% confidence intervals will be computed.
Time Frame: From date of enrollment to death from any cause, assessed up to 2.5 years
Measure: Median (Standard Error); unit: Days
Arm/Group | Treatment (BMS-986205 and Nivolumab)
Number analyzed (Participants) | 8
Days | NA (NA) — Insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: All cause mortality - assessed for up to about 2.5 years. Serious and Other Adverse Events assessed for up to 2 years.
Arm/Group | Treatment (BMS-986205 and Nivolumab)
All-Cause Mortality (participants affected / at risk) | 4/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (BMS-986205 and Nivolumab) (N=8)
Diarrhea (Gastrointestinal disorders) | 1 (1)
AST increase (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (BMS-986205 and Nivolumab) (N=8)
Diarrhea (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 1
Flatulance (Gastrointestinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Maculopapular rash (Skin and subcutaneous tissue disorders) | 2
Alk phos increased (Investigations) | 2
AST increased (Investigations) | 3
ALT increased (Investigations) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Malaise (General disorders) | 1
TSH elevation (Metabolism and nutrition disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT03695250/Prot_SAP_000.pdf